CLINICAL TRIAL: NCT06602427
Title: Shoulder Proprioception: a Comparative Study on Hand Dominance and Sex
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Collaborators: Gamze ÇOBANOĞLU DEMİRKAN (Unknown); Ali ZORLULAR (Unknown); Ahmet GÖKKURT (Unknown); Nihan KAFA (Unknown); Nevin ATALAY GÜZEL (Unknown); Deran OSKAY (Unknown)
Responsible Party: Principal Investigator, Barış SEVEN, Ph.D. research assistant, Gazi University
Other Study IDs: 6
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-08

CONDITIONS: Position Sense; Sex Characteristics; Glenohumeral Joint; Upper Extremity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Shoulder proprioception measurement using isokinetic dynamometer — A Cybex brand isokinetic dynamometer [Cybex NORM®, Humac, CA, USA] was used for shoulder proprioception assessment. Active Joint Position Sensation (AJPS) was evaluated to examine proprioception. AJPS was measured in the sitting position. The target angle was 30° external and 30° internal rotation. The participant was positioned with the elbow in 90° flexion and the wrist in the neutral position. The dynamometer was fixed at 0° to ensure the same starting position for each participant during trials and evaluations. Before starting the test, 3 trials were performed and then the participants were asked to find the target angle 3 times. The amount of error between the target angle and the angle found by the participant was used to describe the accuracy of the AJPS. The arithmetic mean of the result of the 3 tests was recorded for use.

SUMMARY:
The goal of this cross-sectional study is to examine the differences in proprioception sensation depending on sex and dominant side factors in healthy volunteers. Hypothesises:

H0: Shoulder proprioception sensation does not change depending on sex and dominant side factors.

H1: Shoulder proprioception sensation varies depending on sex and dominant side factors.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have agreed to participate in the study after being provided with detailed information about the research will be included in the study.

Exclusion Criteria:

* Individuals who have undergone surgery or experienced trauma in the upper extremity, which impairs hand function, strength, and/or sensation, or who have a fracture or acute orthopedic injury within the last 6 months.
* Individuals with a history of neuromuscular disease, traumatic nerve injury, congenital anomaly, skin infections, or other conditions that could affect the assessment.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy young adults
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2024-09-26 (Actual)

PRIMARY OUTCOMES:
Shoulder proprioception measurement | Participants will be evaluated only once.

CONTACTS AND LOCATIONS:
Locations (1):
- Barış SEVEN, Izmir, Çiğli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No